CLINICAL TRIAL: NCT01843582
Title: A Study to Develop Both a Novel Method for Evaluating the True Size of a Retinal Object on Fundus Photographs and a New Reaction-time Based Method for Studying the Visual Field on Healthy Volunteers
Brief Title: A Study to Determine the Location of the Blind Spot and the Macula-disc Centre Distance on a Fundus Photograph
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T81/2012
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2013-05

CONDITIONS: Generalized Visual Field Contraction or Constriction
Keywords: Keyword: blind spot
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is aimed to develop a new reaction-time based method for examining the visual field and to study the effect of refractive error on the magnification of a fundus photograph in order to evaluate the true size of a retinal feature.

ELIGIBILITY:
Inclusion Criteria:

* No disease that effect the fundus photograph or visual field

Exclusion Criteria:

* any disease that effects the fundus photograph or visual field

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Macula-disc centre distance | one measurement at the start of the study
  Measurement is done on a fundus photograph (one visit and one examination for each patient)

SECONDARY OUTCOMES:
Location of the blind spot | one measurement at the start of the study
  The location of the blind spot is screened using Octopus custom made visual field program at the one visit (one visit and one study for each patient) and a novel reaction-time based visual field device.

CONTACTS AND LOCATIONS:
Overall Officials: Eija Vesti, professor, Study Director — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland